CLINICAL TRIAL: NCT06623136
Title: An Open-label, Multicenter, Single-arm Phase 2 Study of ES102 in Combination With Toripalimab in Subjects With Advanced Non-small Cell Lung Cancer
Brief Title: A Study of ES102 in Combination With Toripalimab in Subjects With Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Elpiscience (Suzhou) Biopharma, Ltd. (Industry)
Responsible Party: Sponsor
Organization: Elpiscience Biopharma, Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES102-2001
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: OX40; PD-1; ES102; JS001; Solid Tumors; INBRX-106
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ES102 in combination with Toripalimab (Experimental)
  Interventions: Drug: ES102; Drug: Toripalimab

INTERVENTIONS:
Drug: ES102 — ES102 is administered via intravenous infusion, once every 21 days.
Drug: Toripalimab — Toripalimab is administered via intravenous infusion, once every 21 days.

SUMMARY:
The aim of this study is to evaluate the efficacy, safety, tolerability, pharmacokinetics (PK) and immunogenicity of ES102 in combination with Toripalimab in subjects with advanced non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Having sufficient understanding of this study and being willing to sign the informed consent form (ICF).
* Males or females, age 18-75 years at the time of signing the informed consent form.
* Histologically or cytologically confirmed, unresectable locally advanced and metastatic non-small cell lung cancer not suitable for radical concurrent chemoradiotherapy.
* Without known EGFR mutation/ALK fusion/ROS1 fusion gene.
* Previous failed concurrent or sequential treatment with systemic platinum-containing chemotherapy and PD-1/PD-L1 inhibitor therapy for NSCLC that cannot be radically resected or not suitable for radical concurrent radio chemotherapy.
* Five consecutive unstained slides from formalin-fixed paraffin-embedded (FFPE) tumor tissue (archived tumor tissue up to 5 years or freshly biopsied tumor tissue) sources are available for PD-L1 testing in the central laboratory.
* PD-L1 TPS ≥50% by 22C3 antibody IHC assay in the central laboratory.
* At least one measurable lesion (in accordance with RECIST v1.1).
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
* Estimated life expectancy of at least 3 months.
* Adequate hematologic, hepatic, renal and coagulation function as defined per protocol.
* Male and female subjects of childbearing potential must be willing to be completely abstinent or to use a highly effective method of contraception (i.e., a failure rate of less than 1%) from the time of signing the informed consent form until 3 months after the last dose of study drug.

Exclusion Criteria:

* Any prior therapy targeting OX40.
* Receipt of any other investigational drug or device intervention within 28 days prior to the first dose of the study drug.
* Receipt of anticancer Chinese herbal therapy within 14 days prior to the first dose of the study drug.
* Receipt of radiotherapy within 14 days prior to the first dose of the study drug.
* Receipt of any other anti-cancer drug(s) including chemotherapy, targeted therapy, immunotherapy, biotherapy, etc., within 28 days or 5 half-lives prior to the first dose of the study drug.
* Prior allogeneic or autologous bone marrow transplant or solid organ transplant.
* The toxicity from prior anti-cancer therapies has not resolved to ≤ Grade 1 per NCI-CTCAE v5.0. Certain exceptions as defined in protocol apply.
* Systemic glucocorticoids (e.g., >10 mg/day of prednisone or equivalent doses of similar drugs) or other immunosuppressive agents were required for systemic treatment within 14 days prior to the first dose of the study drug or during the study period.
* Major surgery within 28 days prior to the first dose of the study drug.
* Receipt of live viral vaccine treatment within 28 days prior to the first dose of the study drug.
* Known allergy to CHO-produced antibodies, which in the opinion of the Investigator suggests an increased potential for hypersensitivity to ES102.
* Subjects with an allergic reaction to the active ingredients ofToripalimab or any of the excipients.
* Known allergy to the pre-medication prescribed in the protocol and unable to receive pre-medication.
* History of invasive malignant tumors other than the study disease within the past two years. Some exceptions as defined per protocol apply.
* History of immune-related adverse events (irAEs) of Grade ≥3 or those that led to discontinuation of treatment. Some exceptions as defined per protocol apply.
* Active autoimmune disease or a known history of autoimmune disease requiring systemic corticosteroid or immunosuppressive treatment.
* Active interstitial lung disease (ILD) or pneumonia; or a history of ILD or (non-infectious) pneumonia requiring corticosteroid or other immunosuppressive treatment.
* Central Nervous System (CNS) metastases.
* Active infection requiring systemic treatment; Human Immunodeficiency Virus (HIV) infection (HIV antibody positive); Hepatitis B Virus (HBV) infection (HBsAg positive) or Hepatitis C Virus (HCV) infection (HCV antibody positive). Some exceptions as defined per protocol apply.
* Cirrhosis, alcoholic hepatitis, drug-induced hepatitis, non-alcoholic steatohepatitis, and hereditary liver diseases.
* History or evidence of cardiovascular abnormalities.
* Pregnant or breastfeeding women.
* Any known, documented, or suspected history of substance abuse that would preclude subject from participation, certain exceptions as defined in protocol apply.
* Any other disease or clinically significant abnormal laboratory parameters that investigator considers may compromise subject safety or study integrity, interfere with subject participation in the trial, or affect the study objectives, including serious medical or psychiatric illness/condition.
* Personnel involved in the design and/or implementation of the study (applicable to sponsor/CRO personnel and site personnel).
* Subjects are unable to comply with the study procedures, restrictions and requirements, in the opinion of Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) assessed by IRC | 1-2 years
  Proportion of subjects achieving complete response (CR) or partial response (PR) according to RECIST v1.1 as assessed by the Independent Review Committee (IRC).

SECONDARY OUTCOMES:
ORR assessed by investigators | 1-2 years
  Proportion of subjects achieving CR or PR according to RECIST v1.1 as assessed by investigators.
Disease control rate (DCR) | 1-2 years
  Proportion of subjects achieving CR, PR or stable disease (SD) according to RECIST v1.1 as assessed by IRC and investigators.
Duration of response (DOR) | 1-2 years
  The time from first documented evidence of CR or PR to disease progression or death, whichever occurs first, in subjects who demonstrate a CR or PR per RECIST v1.1 , as assessed by IRC and investigators.
Progression-free survival (PFS) | 1-2 years
  Time from the date of first study drug administration to disease progression or death, whichever occurs first, as assessed by IRC and investigators.
Overall survival (OS) | 1-2 years
  The time from the date of first study drug administration to the date of death due to any cause.
Adverse events (AE) | 1-2 years
  The number of subjects who experienced an adverse event (AE) will be presented. AE will be collected beginning with subject receiving first dose of the study drug until the time specified in the protocol.
Plasma concentration | 1-2 years
  Plasma concentration will be obtained by laboratory testing of blood samples taken from subjects before and after administration of the study drug.
Immunogenicity Toripalimab | 1-2 years
  Frequency of anti-drug antibodies (ADA) against ES102 or Toripalimab will be determined.

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Cancer Hospital of Shandong First Medical University (Shandong Cancer Institute, Shandong Cancer Hospital), Jinan, Shandong
  - The First Affiliated Hospital of He'nan University of Science and Technology, Luoyang
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - Taizhou Hospital, Taizhou

IPD SHARING:
Plan to Share IPD: No